CLINICAL TRIAL: NCT00967993
Title: A 6-Week Feasibility Trial of a New Formulation of KRX-0502 (Ferric Citrate) in Patients With End-Stage Renal Disease (ESRD)
Brief Title: Trial of a New Formulation of KRX-0502 (Ferric Citrate) in Patients With End-Stage Renal Disease
Status: Completed | Type: Observational
Sponsor: Keryx Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: KRX-0502-202
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-11

CONDITIONS: Hyperphosphatemia; End-stage Renal Disease; Renal Failure Chronic Requiring Hemodialysis
Keywords: hyperphosphatemia; end-stage renal disease; ESRD; hemodialysis; diabetes; dialysis
MeSH Terms: conditions — Hyperphosphatemia; Kidney Failure, Chronic; Diabetes Mellitus | interventions — ferric citrate

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- KRX-0502 (ferric citrate): KRX-0502 will be supplied as one caplet of ferric citrate containing 210 mg of ferric iron as ferric citrate. All patients initiated on study drug will start with a fixed dose of KRX-0502 (ferric citrate) of 6 caplets per day.
  Patients will be titrated at Visits 4, 5, and 6 based on serum phosphorus lab results. If serum phosphorus levels go below normal, there will be a decrease in pills; if serum phosphorus levels go above normal, there wil be an increase in pills. The maximum number of KRX-0502 (ferric citrate) caplets per day will be 12, or 12 g/day of ferric citrate.
  Patients will take study drug orally with meals or snacks or within one hour after their meals or snacks.
  Interventions: Drug: ferric citrate

INTERVENTIONS:
Drug: ferric citrate — KRX-0502 will be supplied as one caplet of ferric citrate containing 210 mg of ferric iron as ferric citrate
  Other Names: KRX-0502

SUMMARY:
The objective of this study is to see if KRX-0502 (ferric citrate) is safe and effective as a dietary phosphate binder in controlling and managing serum phosphorus levels in patients with end-stage renal disease (ESRD).

DETAILED DESCRIPTION:
This is a multi-center, non-blinded, efficacy and tolerability trial in patients with ESRD on dialysis three times per week. Approximately 24 patients (approximately twelve diabetic patients and approximately twelve non-diabetic patients) in Israel will be initiated on KRX-0502 (ferric citrate). The study will consist of a two-week washout period immediately followed by a six-week treatment period in. Patients will be initiated on study drug over two to three weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant, non-lactating females
2. Age > 18 years
3. On thrice weekly hemodialysis for at least the previous three months prior to screening
4. Serum phosphorus levels ≥ 2.5 mg/dL and < 8.5 mg/dL at Screening Visit (Visit 0)
5. Serum phosphorus levels > 5.5 mg/dL at Study Drug Initiation Visit (Visit 3)
6. Taking 3 to 18 tablets/capsules/day of calcium acetate calcium carbonate, lanthanum carbonate, sevelamer (hydrochloride or carbonate), or any combination of these agents as reported by the patient at screening
7. Serum ferritin <1000micrograms/L and Transferrin Saturation (TSAT) <50%
8. Willing to be discontinued from current phosphate binder(s) and initiated on KRX-0502 (ferric citrate)
9. Willing and able to give informed consent

Exclusion Criteria:

1. Parathyroidectomy within six months prior to Screening Visit (Visit 0)
2. Actively symptomatic gastrointestinal bleeding and inflammatory bowel disease
3. Serum phosphorus levels >10.0 mg/dL documented in the three monthly laboratories (done routinely in the dialysis unit) in the three months prior to the Screening Visit (Visit 0)
4. History of multiple drug allergies
5. History of malignancy in the last five years (treated cervical or skin cancer may be permitted if approved by Keryx)
6. Previous intolerance to oral ferric citrate
7. Absolute requirement for oral iron therapy
8. Absolute requirement for Vitamin C (multivitamins [Centrum, Nephrocaps, Renaphro, etc.] allowed)
9. Absolute requirement for calcium, magnesium, or aluminum containing drugs with meals
10. Psychiatric disorder that interferes with the patient's ability to comply with the study protocol
11. Inability to tolerate oral drug intake
12. Planned surgery or hospitalization during the study (scheduled outpatient access surgery allowed)
13. Any other medical condition that renders the patient unable to or unlikely to complete the study or that would interfere with optimal participation in the study or produce significant risk to the patient
14. Receipt of any investigational drug within 30 days of randomization
15. Inability to cooperate with study personnel or history of noncompliance
16. Prior exposure to ferric citrate
17. Patients with hemochromatosis or Thalassemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients selected from pool of dialysis patients at each clinic.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Itamar Raz, MD, Principal Investigator — Hadassah University Hospital-Ein Kerem
Locations (3):
- Israel (3):
  - Barzilai Medical Center Ben-Gurion University, Ashkelon
  - Hadassah University Hospital-Ein Kerem, Jerusalem
  - Assaf Haraofeh Medical Center, Ẕerifin

REFERENCES:
- [Background] Hsu CH, Patel SR, Young EW. New phosphate binding agents: ferric compounds. J Am Soc Nephrol. 1999 Jun;10(6):1274-80. doi: 10.1681/ASN.V1061274. PMID 10361865
- [Background] Yang WC, Yang CS, Hou CC, Wu TH, Young EW, Hsu CH. An open-label, crossover study of a new phosphate-binding agent in haemodialysis patients: ferric citrate. Nephrol Dial Transplant. 2002 Feb;17(2):265-70. doi: 10.1093/ndt/17.2.265. PMID 11812877
- See also: Sponsor Website — http://www.keryx.com

RESULTS

PARTICIPANT FLOW:
Groups:
- KRX-0502: All patients initiated on study drug were started on a fixed dose of KRX-0502 (ferric citrate) of 6 caplets per day. Patients were titrated at Visits 4, 5, and 6 based on serum phosphorus lab results. If serum phosphorus levels went below normal, there was a decrease in pills; if serum phosphorus levels went above normal, there was an increase in pills. The maximum number of KRX-0502 (ferric citrate) caplets per day was 12, or 12 g/day of ferric citrate."
Period: Overall Study
Arm/Group | KRX-0502
Started | 22
Completed | 18
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- KRX-0502: All subjects in this group will receive treatment with KRX-0502, 1g ferric citrate containing approximately 210 mg of ferric iron
Arm/Group | KRX-0502
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (0.8)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15
Region of Enrollment [Number; unit: participants]
  Israel | 22

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome of This Trial Will be the Change in Serum Phosphorus From Baseline to End of Treatment After a Four Week Treatment Period.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- KRX-0502 (Ferric Citrate): Single arm clinical trial of KRX-0502 (ferric citrate)
Arm/Group | KRX-0502 (Ferric Citrate)
Number analyzed (Participants) | 19
mg/dL | -1.53 (1.22)

2. Secondary Outcome: The Incidence of Treatment-emergent Adverse Events (New or Worsened From Study Drug Initiation) Will be Summarized by Body System, Severity, Type of Adverse Event, and Presumed Relationship to the Study Drug.
Time Frame: 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | KRX-0502 (Ferric Citrate)
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 8/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KRX-0502 (Ferric Citrate) (N=22)
Abdominal Pain (Gastrointestinal disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Exacerbation of Constipation (Gastrointestinal disorders) | 1 (1)
Loose Stool Intermittent (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Odor of ferric citrate (Gastrointestinal disorders) | 1 (1)
Clotted A-V Fistula Recurrent (General disorders) | 1 (1)
Exertion Fatigue (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Strange Feeling in Head (General disorders) | 1 (2)
Liver Enzyme Elevation (Hepatobiliary disorders) | 1 (1)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hand Dysaesthsia (Nervous system disorders) | 1 (1)
Decrease in Urea Reduction Rate (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 2 (2)
Rash Diffuse (Skin and subcutaneous tissue disorders) | 1 (1)
Low BP Dizziness Weakness (Vascular disorders) | 1 (1)
Syncope (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No